CLINICAL TRIAL: NCT06284525
Title: Ankle Assistance and Resistance in Older Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northern Arizona University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2137420
Record Dates: First submitted 2024-02-08; First posted 2024-02-29 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Gait training with exoskeleton resistance (Experimental): Participants will complete 20-30 minutes of ankle resistance training on each visit. This will involve walking on a treadmill with stance phase ankle resistance and biofeedback.
  Interventions: Device: Ankle resistance and biofeedback

INTERVENTIONS:
Device: Ankle resistance and biofeedback — An ankle exoskeleton will provide stance phase resistance and a plantar pressure biofeedback system will encourage late stance push-off.

SUMMARY:
The goal of this research protocol is to improve mobility in older individuals through advances in wearable assistive devices by focusing on two specific aims. The first aim is to study if targeted ankle resistance gait training improves walking performance in older individuals. The second aim is to evaluate the potential of wearable assistance at the ankle, knee, and/or hip joints to increase walking performance in older individuals.

DETAILED DESCRIPTION:
The overarching goal of this study is to improve mobility in older adults through advances in wearable assistance (i.e. powered orthoses). This goal will be accomplished by focusing on two specific research aims. The first aim is to study if targeted ankle resistance gait training improves walking performance in older individuals. The second aim is to evaluate the potential of wearable assistance at the ankle, knee, and/or hip joints to increase walking performance in older individuals.

Several powered orthosis conditions will be tested during several modes of walking or running and balance throughout the course of the study. Trials will take place over-ground and/or on a treadmill. Balance trials will take place on a treadmill. Participants will walk for up to 40 minutes. Frequent breaks will be provided between trials and conditions to avoid fatigue; a maximum of 15 minutes of continuous walking will take place between breaks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 85 years old, inclusive.
* Must be able to understand and follow simple directions based on parent report and clinical observation during the history and physical examination.
* Able to provide verbal assent, if appropriate. If the participant is non-verbal, parental interpretation of gesticulation for assent will be used.
* The ability to read and understand English.
* Able to walk at least 30 feet with or without a walking aid
* Able to safely fit into a device configuration and tolerate assistance without knee hyperextension while walking

Exclusion Criteria:

* Any neurological, musculoskeletal or cardiorespiratory injury, health condition ( including pregnancy), or diagnosis that would affect the ability to walk as directed for short periods of time. Note: For elderly participants, a history of joint replacement or joint degeneration that does not impair their ability to walk safely is allowable.
* Participant or parent report that the perspective participant's physician has recommended that they not engage in moderate intensity walking exercise.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gait Training With Exoskeleton Resistance
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: >65 years old
Arm/Group | Gait Training With Exoskeleton Resistance
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in 6MWT
Description: Change (post - baseline) in six minute walk test distance (distance in meters)
Time Frame: Baseline assessment and 1-week post training assessment (at 5 weeks)
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Gait Training With Exoskeleton Resistance
Number analyzed (Participants) | 8
m | 48.3 (50.5)

2. Primary Outcome: Change in Metabolic Power
Description: Change (post - baseline) in metabolic power measured in J/(kgm)
Time Frame: Baseline assessment and 1-week post training assessment (at 5 weeks)
Measure: Mean (Standard Deviation); unit: J/(kgm)
Arm/Group | Gait Training With Exoskeleton Resistance
Number analyzed (Participants) | 8
J/(kgm) | -0.09 (0.58)

3. Primary Outcome: Change in Plantar Flexor Force Production
Description: Change (post - baseline) in manual muscle testing plantar flexor force production measured in N/kg
Time Frame: Baseline assessment and 1-week post training assessment (at 5 weeks)
Measure: Mean (Standard Deviation); unit: N/kg
Arm/Group | Gait Training With Exoskeleton Resistance
Number analyzed (Participants) | 8
N/kg | 0.6 (0.2)

ADVERSE EVENTS:
Time Frame: Approximately 4 weeks
Arm/Group | Gait Training With Exoskeleton Resistance
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT06284525/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT06284525/SAP_001.pdf
  • Informed Consent Form (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT06284525/ICF_002.pdf